CLINICAL TRIAL: NCT02284477
Title: Associations of Exposure to Phthalates With Insulin Resistance and Epigenetic Change
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2014-2075
Record Dates: First submitted 2014-10-30; First posted 2014-11-06 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2014-10

CONDITIONS: Insulin Resistance; Decreased Pulmonary Function
Keywords: Insulin resistance; Pulmonary function; Phthalates
MeSH Terms: conditions — Insulin Resistance; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- non- PVC containing packing materials (Experimental): Participants will be provided food for lunch and dinner with 360mL apple juice which was stored in glass bottle for 24 hours in 4 ℃. After 1 week, participant will cross over to other intervention.
  Interventions: Other: non- PVC containing packing materials
- PVC containing packing materials (Experimental): Participants will be provided food for lunch and dinner with 360mL apple juice which was stored in PVC blood bag for 24 hours in 4 ℃. After 1 week, participant will cross over to other intervention.
  Interventions: Other: PVC containing packing materials
- Only lunch and dinner (No Intervention): Participant received food for lunch and dinner After 1 week, participant get over to each experimental arms.

INTERVENTIONS:
Other: non- PVC containing packing materials — Beverage which was stored in glass bottle for 24 hours in 4 ℃.
  Other Names: Beverage stored in glass bottle
  Arms: non- PVC containing packing materials
Other: PVC containing packing materials — Beverage which was stored in PVC blood bag for 24 hours in 4 ℃.
  Other Names: Beverage stored in blood bag
  Arms: PVC containing packing materials

SUMMARY:
* Phthalate is an endocrine disrupting chemical, which works as an anti-androgenic agent.
* Phthalate is mainly used as PVC plasticizer and easily found in commonly used products such as electronic device, paint, lubricant, surfactant, medical supplies, spray etc. Especially, PVC blood bag used for blood transfusion have been reported to have high level of phthalate concentration.
* Previous studies reported that urinary concentration of phthalate metabolites and HOMA (Homeostatic model assessment, indicator of insulin resistance) has positive association.
* Previous studies also reported negative associations between urinary phthalate concentration and pulmonary function.
* Exposure to phthalates occurs mainly through oral route. Food wrapping with phthalate containing package material is expected to be one of the major contributor for phthalate exposure.
* In this present trial, the investigators are to examine whether increased phthalate exposure by consuming beverage stored in PVC containing packing materials actually effect insulin resistance, pulmonary function and epigenetic feature.
* For this aim, the investigators will conduct a cross-over trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants who understand aim of this study and who provided informed consent

Exclusion Criteria:

* Who did not provided informed consent
* Person who are undergoing or planning to take a treatment due to liver, nervous system, respiratory system, hematologic, oncologic, psychiatric, cardiovascular(angina pectoris, myocardial infarction, stroke etc), endocrinal(Diabetes mellitus, thyroid disease) disorders.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Increase of insulin resistance assessed by HOMA (Homeostatic model assessment) | average 14 hours after consumption of assigned food and beverage

SECONDARY OUTCOMES:
Change of DNA methylation assessed by Percent DNA methylation | average 14 hours after consumption of assigned food and beverage
Decrease of lung function assessed by FEV1 | average 14 hours after consumption of assigned food and beverage
Decrease of lung function assessed by FVC | average 14 hours after consumption of assigned food and beverage
Decrease of lung function assessed by FEV1/FVC | average 14 hours after consumption of assigned food and beverage
Decrease of lung function assessed by FEF25-75 | average 14 hours after consumption of assigned food and beverage
Increased exposure to Phthalate assessed by urinary concentration of metabolites | average 14 hours after consumption of assigned food and beverage

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Chul Hong, MD, PhD, Principal Investigator — College of Medicine, Seoul National Unveirsity
Locations (1):
- Department of Preventive Medicine, College of Medicine, Seoul National University, Seoul, South Korea

REFERENCES:
- [Background] Stahlhut RW, van Wijngaarden E, Dye TD, Cook S, Swan SH. Concentrations of urinary phthalate metabolites are associated with increased waist circumference and insulin resistance in adult U.S. males. Environ Health Perspect. 2007 Jun;115(6):876-82. doi: 10.1289/ehp.9882. Epub 2007 Mar 14. PMID 17589594
- [Background] Rudel RA, Gray JM, Engel CL, Rawsthorne TW, Dodson RE, Ackerman JM, Rizzo J, Nudelman JL, Brody JG. Food packaging and bisphenol A and bis(2-ethyhexyl) phthalate exposure: findings from a dietary intervention. Environ Health Perspect. 2011 Jul;119(7):914-20. doi: 10.1289/ehp.1003170. Epub 2011 Mar 30. PMID 21450549
- [Background] Singh S, Li SS. Epigenetic effects of environmental chemicals bisphenol A and phthalates. Int J Mol Sci. 2012;13(8):10143-10153. doi: 10.3390/ijms130810143. Epub 2012 Aug 15. PMID 22949852
- [Background] Manikkam M, Tracey R, Guerrero-Bosagna C, Skinner MK. Plastics derived endocrine disruptors (BPA, DEHP and DBP) induce epigenetic transgenerational inheritance of obesity, reproductive disease and sperm epimutations. PLoS One. 2013;8(1):e55387. doi: 10.1371/journal.pone.0055387. Epub 2013 Jan 24. PMID 23359474
- [Background] Kim JH, Hong YC. HSP70-hom gene polymorphisms modify the association of diethylhexyl phthalates with insulin resistance. Environ Mol Mutagen. 2014 Dec;55(9):727-34. doi: 10.1002/em.21884. Epub 2014 Jul 7. PMID 25044062
- [Background] Kim JH, Park HY, Bae S, Lim YH, Hong YC. Diethylhexyl phthalates is associated with insulin resistance via oxidative stress in the elderly: a panel study. PLoS One. 2013 Aug 19;8(8):e71392. doi: 10.1371/journal.pone.0071392. eCollection 2013. PMID 23977034
- [Background] Hoppin JA, Tolbert PE, Flagg EW, Blair A, Zahm SH. Use of a life events calendar approach to elicit occupational history from farmers. Am J Ind Med. 1998 Nov;34(5):470-6. doi: 10.1002/(sici)1097-0274(199811)34:53.0.co;2-u. PMID 9787851
- [Background] Zahm SH, Colt JS, Engel LS, Keifer MC, Alvarado AJ, Burau K, Butterfield P, Caldera S, Cooper SP, Garcia D, Hanis C, Hendrikson E, Heyer N, Hunt LM, Krauska M, MacNaughton N, McDonnell CJ, Mills PK, Mull LD, Nordstrom DL, Outterson B, Slesinger DP, Smith MA, Stallones L, Stephens C, Sweeney A, Sweitzer K, Vernon SW, Blair A. Development of a life events/icon calendar questionnaire to ascertain occupational histories and other characteristics of migrant farmworkers. Am J Ind Med. 2001 Nov;40(5):490-501. doi: 10.1002/ajim.1117. PMID 11675618
- [Background] van der Mei IA, Blizzard L, Ponsonby AL, Dwyer T. Validity and reliability of adult recall of past sun exposure in a case-control study of multiple sclerosis. Cancer Epidemiol Biomarkers Prev. 2006 Aug;15(8):1538-44. doi: 10.1158/1055-9965.EPI-05-0969. PMID 16896046